CLINICAL TRIAL: NCT01587339
Title: Systematic Review: Retigabine for Adjunctive Therapy in Partial Epilepsy
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115049
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — ezogabine; Lacosamide; Zonisamide; Pregabalin; eslicarbazepine; eslicarbazepine acetate

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Drug-resistant (or refractory) partial epilepsy of all types: Drug-resistant (or refractory) partial epilepsy of all types
  Interventions: Drug: retigabine/ezogabine; Drug: lacosamide; Drug: zonisamide; Drug: pregabalin; Drug: eslicarbazepine

INTERVENTIONS:
Drug: retigabine/ezogabine — oral - all doses
  Other Names: Trobalt (R); Potiga (R)
Drug: lacosamide — oral - all doses
  Other Names: Vimpat
Drug: zonisamide — oral - all doses
  Other Names: Zonegran
Drug: pregabalin — oral - all doses
  Other Names: Lyrica
Drug: eslicarbazepine — oral - all doses
  Other Names: Zebinix

SUMMARY:
There are a number of anti-epileptic drugs available for the treatment of partial onset seizures in patients with epilepsy. This study is a systematic review of the published literature on anti-epileptic drugs and is designed to compare the relative effectiveness and tolerability of a selection of them with retigabine. The drugs chosen for this comparison were lacosamide, pregabalin, tiagabine, zonisamide and eslicarbazepine. They were chosen because they belong to the newer generation of drugs for epilepsy (as does retigabine) and they have a similar license as well as having published data from studies that were conducted in similar patient populations with similar methods. GSK commissioned YHEC (York Health Economic Consortium) to carry out this review and analysis. YHEC identified relevant studies from international databases. These studies had compared one of the chosen anti-epileptic drugs with placebo. The results were pooled and combined in order to summarize the data for individual drugs as well to compare the results for different drugs with each other and with retigabine. Since none of the individual clinical studies compared one active drug with another, this systematic review is an indirect comparison of these drugs, using an established and recognised methodology which has well understood limitations.

ELIGIBILITY:
Inclusion Criteria:

* Have participated to a study that meets the following criteria:
* Be a study of retigabine, eslicarbazepine, lacosamide, zonisamide, pregabalin or tiagabine as an adjuvant therapy, compared to placebo or another drug;
* Be a randomized, placebo-controlled, add-on trial, or a parallel trial or cross-over trial in which data from the first treatment period could be treated as a parallel study;
* Have recruited patients with drug-resistant partial epilepsy (i.e., simple partial, complex partial, and/or secondarily generalised tonic-clonic seizures not controlled by at least 1 or more other AEDs);
* Have a maintenance treatment period of 8 weeks or longer, with a prospective baseline of minimum 4 weeks.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We included published papers on studies that had recruited drug-resistant (or refractory) partial epilepsy of all types
Sampling Method: Non-Probability Sample
Enrollment: 6498 (Actual)
Dates: Start 2010-09; Primary Completion 2011-03 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Responder Rate | Duration of studies included in the systematic review up to 28 weeks of double blind period
  Proportion of patients who respond to treatment (50% reduction in seizure frequency from baseline)
Median Seizure reduction | Duration of studies included in the systematic review up to 28 weeks of double blind period
  Median percent reduction in seizure frequency from baseline
Seizure severity | Duration of studies included in the systematic review up to 28 weeks of double blind period
  Seizure severity (any definitions acceptable)
Time to onset of treatment effect | Duration of studies included in the systematic review up to 28 weeks of double blind period
  Time to onset of treatment effect
Seizure free patients | Duration of studies included in the systematic review up to 28 weeks of double blind period
  Proportion of patients who are seizure free (and time period over which this was measured)
Changes in HRQoL | Duration of studies included in the systematic review up to 28 weeks of double blind period
  Changes in HRQoL
All drop outs | Duration of studies included in the systematic review up to 28 weeks of double blind period
  Proportion of patients who drop out of the studies for any reason
Drop outs due to AE | Duration of studies included in the systematic review up to 28 weeks of double blind period
  Proportion of patients who drop out of the studies (as a result of adverse events i.e. tolerability)
Adverse events | Duration of studies included in the systematic review up to 28 weeks of double blind period
  Percentage of patients reporting 5 key adverse events identified by the Cochrane Epilepsy Group as common and important adverse effects of antiepileptic drugs: ataxia, dizziness, fatigue, nausea or somnolence
Mortality | Duration of studies included in the systematic review up to 28 weeks of double blind period
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] Martyn-St James M, Glanville J, McCool R, Duffy S, Cooper J, Hugel P, Lane PW. The efficacy and safety of retigabine and other adjunctive treatments for refractory partial epilepsy: a systematic review and indirect comparison. Seizure. 2012 Nov;21(9):665-78. doi: 10.1016/j.seizure.2012.07.011. Epub 2012 Aug 14. PMID 22902288